CLINICAL TRIAL: NCT01791387
Title: Dovitinib In 1st-Line Renal Cell Carcinoma, an Investigation Into Tumour GENe Status and Correlation With Efficacy - 1st Exploratory Study
Brief Title: 1st-line Activity of Dovitinib and Correlation With Genetic Changes in RCC
Acronym: DILIGENCE-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Auckland District Health Board (Other Government)
Collaborators: University of Auckland, New Zealand (Other); IGENZ, Ltd., Auckland (Unknown); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258AAU02T; ACTRN12612000140853 (Registry Identifier: Australian Clinical Trials Registry)
Record Dates: First submitted 2013-01-08; First posted 2013-02-15 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: Renal cell; Kidney; Cancer; Metastatic carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Carcinoma | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dovitinib (Experimental): Dovitinib 500 mg taken orally once daily 5 days on / 2 days off, until disease progression
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib — Patients will be treated with dovitinib (500 mg orally, once daily 5 days on/2 days off) until disease progression, intolerability, patient refusal, death or study drug discontinuation for any other reason. Dovitinib should be ingested at least 1 hour prior to a meal or at least 2 hours following a meal at approximately the same time each day.
  If patients cannot tolerate the protocol-specified dosing schedule, dose reductions or treatment interruptions are permitted. When necessary, dovitinib may be reduced to 400 mg for 5 days on/2 days off. If an additional dose reduction is required, dovitinib may be reduced to 300 mg dose 5 days on/2 days off. Once dose is reduced due to an adverse event, it cannot be re-escalated. Patients are allowed only 2 dose reductions.
  Other Names: TKI258

SUMMARY:
The main purpose of this study is to find out how useful dovitinib is when given as the initial treatment to participants with advanced kidney cancer, that has spread to other parts of the body. The usefulness of dovitinib will be assessed by: how long the disease is controlled while participants are receiving the drug, the proportion of participants who get a reduction in the size of their tumours and how long participants live (both while on dovitinib and on any subsequent therapy they may receive).

If participants have secondary disease in the bones, the study will evaluate how useful dovitinib is in controlling this site of disease. In addition, this study will look for changes in the genetic makeup of tumour cells and see if some of these changes are associated with a benefit from dovitinib. The study will also compare and contrast the genetic changes in the primary tumour cells with cells from secondary tumour specimens, and with cells from tumour specimens taken if a participant's disease has worsened. The purpose of the latter is to identify possible ways in which the tumour becomes resistant to the study drug.

DETAILED DESCRIPTION:
The purpose of this prospective, single centre, non-randomised, open-label, phase II study will evaluate the activity of dovitinib in the treatment naïve population of patients with advanced RCC.

Background: Prior to the middle of last decade, the only systemic therapy for patients with advanced RCC was immunotherapy (interleukin-2 and interferon-alpha) with limited effectiveness and a multitude of side-effects. Since 2006, there have been 6 targeted therapies that have been FDA-registered for the treatment of advanced RCC; the anti-VEGFR tyrosine kinase inhibitors (sunitinib, sorafenib and pazopanib), the anti-VEGF antibody bevacizumab (with interferon-alpha) and the mTOR inhibitors (everolimus and temsirolimus). These treatments have significantly advanced outcomes for patients with this disease but unfortunately they do not represent cures. The median overall survival for patients treated with a standard first-line therapy (sunitinib) is just over 2 years and the median PFS for subjects receiving this agent is only 11 months. This means that the typical time it takes for subjects to develop resistance to standard first-line tyrosine kinase inhibitor (TKI) treatment, as evidenced by significant tumour growth on imaging, is under 1 year.

Despite the recent rapid advancements in the treatment options for subjects with advanced RCC, there is still an unmet need for more effective therapeutic options for patients with this disease so as to improve survival and make steps towards the ultimate treatment aim for patients with metastatic disease - cure. Available data suggests that dovitinib is a very active agent in metastatic RCC. If it has efficacy in the heavily pre-treated RCC population, one would expect it to be considerably more active when it is moved forward into the first-line setting.

Dovitinib is a broad-targeted receptor Tyrosine Kinase Inhibitor (TKI) primarily active against three receptors that mediate tumour growth and survival: vascular endothelial growth factor receptor (VEGFR), platelet-derived growth factor receptor (PDGFR) and fibroblast growth factor receptor (FGFR). A distinguishing feature of dovitinib (compared to other anti-VEGFR TKI's) is its FGFR inhibition. Up-regulation of the fibroblast growth factor receptor 1 (FGFR1) pathway has been demonstrated in metastatic RCC and is a postulated mechanism of resistance to anti-VEGFR therapies. This is thought to be one of the reasons why dovitinib has activity in subjects treated with prior anti-VEGFR therapies. If we move the FGFR inhibition forward into the first-line setting (by using dovitinib) we hope to be able prevent or delay the development of resistance acquired through FGFR up-regulation. We hope this may allow subjects to remain on first-line therapy for much longer and in doing so improve survival and outcomes for this group of patients.

Dovitinib has been studied in heavily pre-treated subjects with metastatic RCC, and in these phase I/II studies it looks very active. If it has efficacy in the heavily pre-treated RCC population, it is possible it would be more active when it is moved forward in to the first-line setting.

While we have good prognostic markers to risk-stratify subjects with RCC, there is a lack of predictive markers to guide us as to which patients are best served with each of the different agents available for use. It is therefore imperative that drug development studies in this disease have companion biomarker analysis to identify potentially useful predictive biomarkers for future research. This study also aims to explore (using FISH) the amplification/deletion status of range of genes-of-interest, selected for their relevance to the biology of RCC and the mechanism-of-action of dovitinib. Amplification/deletion of these genes will be further validated using DNA sequencing. The status of these genes-of-interest will be correlated with outcomes of these subjects treated with dovitinib.

The hypothesis of this study is that dovitinib will demonstrate anti-tumour activity when administered to subjects with advanced RCC in the first-line setting and that this activity will correlate with FGFR gene amplification status.

The primary objective is to evaluate the activity of dovitinib in the treatment naïve population of patients with advanced RCC.

Secondary Objectives:

* To determine the gene amplification status for FGFR-1,-2,-3 in this patient population
* To measure the strength of the correlation between measures of clinical efficacy and FGFR gene amplification status
* To further evaluate safety

Exploratory Objectives:

* To assess for amplifications/deletions for genes related to RCC biology in this group of subjects treated with dovitinib.
* To correlate gene amplification status with DNA gene sequence.
* To evaluate differences in tumour gene status between primary and metastatic samples from same subject and again on post-treatment biopsy to elucidate mechanisms of resistance to dovitinib.
* To evaluate effects of dovitinib on bone metastases and pain.

Investigational treatment: Thirty patients from the greater Auckland region will be treated with dovitinib (500 mg p.o. o.d., 5 days on/2 days off) until disease progression, unacceptable toxicity, patient withdrawal or death.

The primary analysis will be performed when 20 progression and/or death events have occurred. No interim efficacy analysis is planned for this study. However, an independent Data Monitoring Committee (DMC) will review data collection (including analysing the adverse event information) and will meet at specified time points during the study.

Visit schedule: Patients will attend clinic visits every 3 weeks while on treatment. Tumour response assessments will occur every 9 weeks until week 54, then every 12 weeks thereafter until disease progression (estimated median time to disease progression = 16 months). Once all patients have completed study treatment, patients will continue to be followed up 3-monthly until approximately 2 months after 20 death events have occurred.

For each patient there will be three separate phases in the study: pre-treatment (screening & baseline), treatment and follow-up.

Pre-treatment phase (Screening/Baseline): The patient must provide a signed informed consent form (ICF) prior to any study related procedure. A screening period of 28 days is allowed to assess eligibility. Radiologic evaluation (CT of the head, chest, abdomen and pelvis) and baseline tumour measurement using RECIST v1.1 will be performed. Other screening and baseline assessments include ECG & echocardiogram to assess cardiac function, performance status assessment (ECOG & WHO), physical examination (including the buccal cavity), height, weight & vital signs. Laboratory investigations include haematology, chemistry, amylase, lipase, serum lipid profile, coagulation, urinalysis, thyroid function, cardiac enzymes and pregnancy test (if applicable). Disease specific information, general medical information including medical history, concomitant medications, prognostic group according to Heng criteria and demographic data will also be collected.

Treatment phase: This study does not have a fixed treatment duration, as patients will continue therapy until disease progression, intolerable toxicity or withdrawal. Following study inclusion and initiation of study treatment, the patient should visit the site on day 1, 8 and 15 during cycle 1, then day 1 of every subsequent cycle. Patients will have their first dose of study treatment on Day 1, Cycle 1. A study cycle is defined as a period of 21 days.

Tumour response will be evaluated every 3 cycles after registration until week 54, then every 4 cycles until documented disease progression. ECOG performance status will be assessed on day 1 of every cycle. Safety assessments are routinely performed including collection of adverse events (AEs), Serious Adverse Events (SAEs), concomitant medications, vital signs, physical examination, weight, haematological and biochemistry assessments, urinalysis, thyroid function and cardiac enzymes. ECG, amylase, lipase, serum lipids and coagulation will be measured if clinically indicated. An echocardiogram will be performed at weeks 12 and 24, and as clinically indicated. Plasma for storage will be collected on Day 1 of Cycles 1 and 3. Participants with bone metastases will have plasma collected for C-telopeptide testing on day 1 of weeks 1, 2 and 13, and will complete a Quality of Life questionnaire (FACT-BP) at 4 time points: on day 1 of weeks1, 2, 4 and 13.

The End of Treatment (EOT) visit will take place approximately 7 days after the last dose of dovitinib. At this visit the following assessments will be performed and the following data collected: physical examination, ECOG performance status, weight, vital signs, adverse events, concomitant medications, antineoplastic therapies, haematology, biochemistry, amylase and lipase measurements.

Safety follow-up: All patients who discontinue study treatment will have a safety follow-up visit within 30 days of the last dose of dovitinib. Safety assessments will include collection of AEs, SAEs, vital signs, concomitant medications and any new antineoplastic therapies. Patients who progress will be invited to provide an (optional) additional biopsy sample of their tumour, at least 10 days after the last dose of dovitinib, but before any new anticancer therapies are initiated.

Efficacy follow-up: Patients who discontinue the study treatment for reasons other than progression will continue to have radiologic assessments, using the same schedule as for patients who remain on treatment, until documented disease progression.

Survival follow-up: Patients who have discontinued study treatment will be followed-up for survival every 3 months by clinical visits or telephone call until death occurs, the patient is lost to follow-up, or withdraws consent for follow-up for survival. Further treatment will be at the discretion of the investigator.

Statistical Methods: All data will be presented descriptively as means, medians or proportions. Progression free and overall survival from the first dose of dovitinib until disease progression or death will be determined using the method of Kaplan-Meier. The correlation between PFS, OS and baseline biomarker status as well as FGFR gene amplification status will be measured using Spearman's rho. Generalized estimating equations (GEE) for repeated measures will also be used to test the significance of changes in biomarker amplification status relative to baseline. Ordinal logistic regression analysis using a repeated measures structure will be applied to compare bone pain control over the treatment period relative to baseline.

Sample Size Calculation and Expected Duration: The response rate (RR) reported for sunitinib, when studied in a phase III trial versus interferon in the first-line setting was approximately 31%, with a 95%CI ranging from 26 to 36% (Motzer, NEJM 356: 115, 2007). The target sample size in this phase II study is 30, which was based on the assumption that the RR for dovitinib would fall within the range of sunitinib. With such a sample size, the prevalence of dovitinib RR using RECIST 1.1 will be measured with a precision that extends to 15 percentage points, with a 95% probability.

ELIGIBILITY:
Inclusion Criteria:

* Advanced renal cell (clear cell) carcinoma confirmed histologically, including either distant metastases or locally advanced disease that is not resectable or potentially resectable following response. Sarcomatoid change is allowed if clear cell predominant. Histological variants, papillary, chromophobe and collecting duct carcinoma are not allowed.
* Availability of FFPE tissue for gene status analysis. If unavailable, an image-guided biopsy of a metastatic disease site is required.
* Evaluable disease by RECIST 1.1 criteria
* ECOG (WHO) performance status 0 or 1
* Age ≥ 18 years
* Absolute neutrophil count ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L; haemoglobin > 9 g/dL; serum total bilirubin ≤ 1.5 x ULN; ALT and AST ≤ 3.0 x ULN; serum creatinine ≤ 1.5 x ULN or creatinine clearance >35 ml/min by Cockcroft and Gault.

Exclusion Criteria:

* Uncontrolled brain metastases. For know brain metastases, definitive treatment with either surgery, stereotactic radiotherapy or whole brain radiotherapy is required. Patients must be neurologically stable for > 4 weeks after CNS treatment ends, and either be off corticosteroids or receiving a low daily dose.
* Another primary malignancy within 3 years prior to starting study treatment, except for adequately treated basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, or in-situ carcinoma of the uterine cervix. If another primary tumour was noted within this period, a metastatic disease site biopsy is required to confirm renal origin.
* Prior systemic anticancer treatment for renal carcinoma. Prior bisphosphonates are allowed.
* Radiotherapy ≤ 4 weeks prior to starting the study drug or non-recovery from related toxicities. Palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting study drug is allowed.
* Major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic) ≤ 4 weeks prior to starting study treatment or non-recovery from surgical side effects.
* History of pulmonary embolism or untreated deep venous thrombosis within the past 6 months. If a history of PE or DVT within the past 6 months is present, patients must be clinically stable on appropriate doses of anticoagulation as per thrombosis specialist advice.
* Impaired cardiac function or clinically significant cardiac diseases, including history of serious uncontrolled ventricular arrhythmias; clinically significant resting bradycardia; LVEF assessed by 2-D echocardiogram < 50% or lower limit of normal (whichever is higher) or multiple gated acquisition scan < 45% or lower limit of normal (whichever is higher). Within 6 months prior to starting study drug: myocardial infarction, severe/unstable angina, coronary artery bypass graft, congestive heart failure, cerebrovascular accident, transient ischemic attack; uncontrolled hypertension defined by a SBP ≥ 160 mm Hg and/or DBP ≥ 90 mm Hg, with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication is allowed before study entry.
* Impaired gastrointestinal function or GI disease that may significantly alter dovitinib absorption, e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome, or small bowel resection.
* Cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Known diagnosis of human immunodeficiency virus infection (testing is not mandatory)
* Current full dose anticoagulation treatment with therapeutic doses of warfarin, dabigatran or anti-platelet therapy. Treatment with ≤ 100mg acetylsalicyclic acid daily is allowed as are therapeutic or prophylactic doses of low molecular weight heparin, provided there is no recent evidence of bleeding.
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. infection, diabetes) that could cause unacceptable safety risks or compromise protocol compliance.
* Pregnant or breast-feeding women
* Women of child-bearing potential or fertile males not using effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) as assessed by RECIST 1.1. | From baseline until documented disease progression, estimated to be up to 65 weeks
  Description: Subjects will undergo baseline radiology assessment with a CT scan of the chest, abdomen, pelvis and head within 4 weeks of registration. Thereafter subjects will then undergo CT scans of the chest, abdomen and pelvis (where possible using the same technique) every 9 weeks until week 54. From week 54 onward, subjects will undergo CT scans of the chest, abdomen and pelvis every 12 weeks until disease progression. Tumour responses will be evaluated using RECIST 1.1. Confirmation of responses (PR/CR) with repeat CT is not required as the primary end-point is PFS. CT will be the only imaging modality required for subjects on study. The RECIST 1.1 assessments will be done in Auckland by one of the members of the Tumour Response EvAluation Team (TREAT) who have expertise in RECIST reporting.

SECONDARY OUTCOMES:
Response rate (RR) using RECIST 1.1. | Change from baseline until disease progression, estimated to be up to 65 weeks
  Assessed every 9 weeks until week 54, then every 12 weeks until disease progression.
Proportion of subjects who are FGFR-1,-2,-3 amplified using gene analysis by Fluorescent in-situ hybridization | Baseline
Efficacy (PFS, RR, OS) by FGFR gene amplification status as measured by Spearman's rho correlation coefficient | Baseline until documented disease progression, estimated to be up to 65 weeks
  Assessed every 9 weeks until week 54, then every 12 weeks until disease progression.
Safety profile of dovitinib (specifically in this first-line patient population) using NCI CTCAE v4.0 | 8 months
  Also assessed at 12 and 24 months
Safety profile of dovitinib (specifically in this first-line patient population) using NCI CTCAE v4.0 | Baseline until documented disease progression, estimated to be up to 65 weeks
  Assessed weekly for weeks 1-3, then every 3 weeks until disease progression.
Proportion of subjects who are FGFR-1,-2,-3 amplified using gene analysis by Fluorescent in-situ hybridization | Disease progression, estimated to be up to 65 weeks.
  Also assessed at 8 and 24 months
Safety profile of dovitinib (specifically in this first-line patient population) using NCI CTCAE v4.0 | 12 months
Safety profile of dovitinib (specifically in this first-line patient population) using NCI CTCAE v4.0 | 24 months
  Also assessed at 8 and 12 months
Safety profile of dovitinib (specifically in this first-line patient population) using NCI CTCAE v4.0 | From documented disease progression up to 2 years.
  Assessed 3-monthly for up to 2 years

OTHER OUTCOMES:
Exploratory objective outcome: Assessment of gene amplifications/deletions related to RCC biology | Baseline
  Proportion of subjects whose tumours have deletion of; VHL, FHIT, PTEN and amplification of; PI3KCA, AKT, MYC, EGFR, PDGFR/CSF-1R, PDGF, imbalance of 1p1q and the correlation of the gene status with clinical outcomes
Exploratory objective outcome: Correlation of gene amplification status with DNA gene sequence | Baseline
  • Correlation between gene amplification status by FISH and DNA sequence using SequenomTM, OncoCartaTM Panel v 1.0
Exploratory objective outcome: Evaluation of differences in tumour gene status between primary and metastatic samples from same subject and again on post-treatment biopsy to elucidate mechanisms of resistance to dovitinib | Baseline
  Discordance in genes-of-interest between and primary and metastatic tumour samples as well as with post-study tumour biopsy (upon progression)
Exploratory endpoint outcome: Effects of dovitinib on bone metastases and pain | Change from baseline until week 1
  Change in FACT-BP score, CTX levels and opioid usage in subjects with bone metastases. Also assessed at week 13.
Exploratory objective outcome: Assessment of gene amplifications/deletions related to RCC biology | Disease progression, estimated to be up to 65 weeks
  Proportion of subjects whose tumours have deletion of; VHL, FHIT, PTEN and amplification of; PI3KCA, AKT, MYC, EGFR, PDGFR/CSF-1R, PDGF, imbalance of 1p1q and the correlation of the gene status with clinical outcomes
Exploratory objective outcome: Correlation of gene amplification status with DNA gene sequence | Disease progression, estimated to be up to 65 weeks
  • Correlation between gene amplification status by FISH and DNA sequence using SequenomTM, OncoCartaTM Panel v 1.0
Exploratory objective outcome: Evaluation of differences in tumour gene status between primary and metastatic samples from same subject and again on post-treatment biopsy to elucidate mechanisms of resistance to dovitinib | Disease progression, estimated to be up to 65 weeks
  Discordance in genes-of-interest between and primary and metastatic tumour samples as well as with post-study tumour biopsy (upon progression)
Exploratory endpoint outcome: Effects of dovitinib on bone metastases and pain | Change from baseline until week 13
  Change in FACT-BP score, CTX levels and opioid usage in subjects with bone metastases. Also assessed at week 1.

CONTACTS AND LOCATIONS:
Overall Officials: Reuben Broom, MBChB, FRACP, Study Chair — Auckland Hospital
Locations (1):
- Auckland Hospital, Auckland, New Zealand

REFERENCES:
- [Background] Gupta K, Miller JD, Li JZ, Russell MW, Charbonneau C. Epidemiologic and socioeconomic burden of metastatic renal cell carcinoma (mRCC): a literature review. Cancer Treat Rev. 2008 May;34(3):193-205. doi: 10.1016/j.ctrv.2007.12.001. Epub 2008 Mar 4. PMID 18313224
- [Background] Chow WH, Devesa SS, Warren JL, Fraumeni JF Jr. Rising incidence of renal cell cancer in the United States. JAMA. 1999 May 5;281(17):1628-31. doi: 10.1001/jama.281.17.1628. PMID 10235157
- [Background] Hollingsworth JM, Miller DC, Daignault S, Hollenbeck BK. Five-year survival after surgical treatment for kidney cancer: a population-based competing risk analysis. Cancer. 2007 May 1;109(9):1763-8. doi: 10.1002/cncr.22600. PMID 17351954
- [Background] Motzer RJ, Hutson TE, Tomczak P, Michaelson MD, Bukowski RM, Oudard S, Negrier S, Szczylik C, Pili R, Bjarnason GA, Garcia-del-Muro X, Sosman JA, Solska E, Wilding G, Thompson JA, Kim ST, Chen I, Huang X, Figlin RA. Overall survival and updated results for sunitinib compared with interferon alfa in patients with metastatic renal cell carcinoma. J Clin Oncol. 2009 Aug 1;27(22):3584-90. doi: 10.1200/JCO.2008.20.1293. Epub 2009 Jun 1. PMID 19487381
- [Background] Sibilia M, Fleischmann A, Behrens A, Stingl L, Carroll J, Watt FM, Schlessinger J, Wagner EF. The EGF receptor provides an essential survival signal for SOS-dependent skin tumor development. Cell. 2000 Jul 21;102(2):211-20. doi: 10.1016/s0092-8674(00)00026-x. PMID 10943841
- [Background] Arteaga CL. The epidermal growth factor receptor: from mutant oncogene in nonhuman cancers to therapeutic target in human neoplasia. J Clin Oncol. 2001 Sep 15;19(18 Suppl):32S-40S. PMID 11560969
- [Background] Cohen P. Protein kinases--the major drug targets of the twenty-first century? Nat Rev Drug Discov. 2002 Apr;1(4):309-15. doi: 10.1038/nrd773. PMID 12120282
- [Background] Collett MS, Erikson RL. Protein kinase activity associated with the avian sarcoma virus src gene product. Proc Natl Acad Sci U S A. 1978 Apr;75(4):2021-4. doi: 10.1073/pnas.75.4.2021. PMID 205879
- [Background] Takahashi Y, Kitadai Y, Bucana CD, Cleary KR, Ellis LM. Expression of vascular endothelial growth factor and its receptor, KDR, correlates with vascularity, metastasis, and proliferation of human colon cancer. Cancer Res. 1995 Sep 15;55(18):3964-8. PMID 7664263
- [Background] Mizuki M, Fenski R, Halfter H, Matsumura I, Schmidt R, Muller C, Gruning W, Kratz-Albers K, Serve S, Steur C, Buchner T, Kienast J, Kanakura Y, Berdel WE, Serve H. Flt3 mutations from patients with acute myeloid leukemia induce transformation of 32D cells mediated by the Ras and STAT5 pathways. Blood. 2000 Dec 1;96(12):3907-14. PMID 11090077
- [Background] Deininger MW, Goldman JM, Melo JV. The molecular biology of chronic myeloid leukemia. Blood. 2000 Nov 15;96(10):3343-56. No abstract available. PMID 11071626
- [Background] Dvorak HF. Rous-Whipple Award Lecture. How tumors make bad blood vessels and stroma. Am J Pathol. 2003 Jun;162(6):1747-57. doi: 10.1016/s0002-9440(10)64309-x. No abstract available. PMID 12759232
- [Background] Auguste P, Javerzat S, Bikfalvi A. Regulation of vascular development by fibroblast growth factors. Cell Tissue Res. 2003 Oct;314(1):157-66. doi: 10.1007/s00441-003-0750-0. Epub 2003 Jul 8. PMID 12851809
- [Background] Casanovas O, Hicklin DJ, Bergers G, Hanahan D. Drug resistance by evasion of antiangiogenic targeting of VEGF signaling in late-stage pancreatic islet tumors. Cancer Cell. 2005 Oct;8(4):299-309. doi: 10.1016/j.ccr.2005.09.005. PMID 16226705
- [Background] Bergers G, Song S, Meyer-Morse N, Bergsland E, Hanahan D. Benefits of targeting both pericytes and endothelial cells in the tumor vasculature with kinase inhibitors. J Clin Invest. 2003 May;111(9):1287-95. doi: 10.1172/JCI17929. PMID 12727920
- [Background] Zhang W, Stoica G, Tasca SI, Kelly KA, Meininger CJ. Modulation of tumor angiogenesis by stem cell factor. Cancer Res. 2000 Dec 1;60(23):6757-62. PMID 11118063
- [Background] Dowlati A, Haaga J, Remick SC, Spiro TP, Gerson SL, Liu L, Berger SJ, Berger NA, Willson JK. Sequential tumor biopsies in early phase clinical trials of anticancer agents for pharmacodynamic evaluation. Clin Cancer Res. 2001 Oct;7(10):2971-6. PMID 11595684
- [Background] Wolff AC, Hammond ME, Schwartz JN, Hagerty KL, Allred DC, Cote RJ, Dowsett M, Fitzgibbons PL, Hanna WM, Langer A, McShane LM, Paik S, Pegram MD, Perez EA, Press MF, Rhodes A, Sturgeon C, Taube SE, Tubbs R, Vance GH, van de Vijver M, Wheeler TM, Hayes DF; American Society of Clinical Oncology/College of American Pathologists. American Society of Clinical Oncology/College of American Pathologists guideline recommendations for human epidermal growth factor receptor 2 testing in breast cancer. Arch Pathol Lab Med. 2007;131(1):18-43. doi: 10.5858/2007-131-18-ASOCCO. PMID 19548375
- [Background] Tsimafeyeu I, Demidov L, Stepanova E, Wynn N, Ta H. Overexpression of fibroblast growth factor receptors FGFR1 and FGFR2 in renal cell carcinoma. Scand J Urol Nephrol. 2011 Apr;45(3):190-5. doi: 10.3109/00365599.2011.552436. Epub 2011 Feb 18. PMID 21329481
- [Background] Rini BI. Metastatic renal cell carcinoma: many treatment options, one patient. J Clin Oncol. 2009 Jul 1;27(19):3225-34. doi: 10.1200/JCO.2008.19.9836. Epub 2009 May 26. PMID 19470934
- [Background] Gronwald J, Storkel S, Holtgreve-Grez H, Hadaczek P, Brinkschmidt C, Jauch A, Lubinski J, Cremer T. Comparison of DNA gains and losses in primary renal clear cell carcinomas and metastatic sites: importance of 1q and 3p copy number changes in metastatic events. Cancer Res. 1997 Feb 1;57(3):481-7. PMID 9012478
- [Background] Velickovic M, Delahunt B, Storkel S, Grebem SK. VHL and FHIT locus loss of heterozygosity is common in all renal cancer morphotypes but differs in pattern and prognostic significance. Cancer Res. 2001 Jun 15;61(12):4815-9. PMID 11406557
- [Background] Meric-Bernstam F, Gonzalez-Angulo AM. Targeting the mTOR signaling network for cancer therapy. J Clin Oncol. 2009 May 1;27(13):2278-87. doi: 10.1200/JCO.2008.20.0766. Epub 2009 Mar 30. PMID 19332717
- [Background] Chen M, Ye Y, Yang H, Tamboli P, Matin S, Tannir NM, Wood CG, Gu J, Wu X. Genome-wide profiling of chromosomal alterations in renal cell carcinoma using high-density single nucleotide polymorphism arrays. Int J Cancer. 2009 Nov 15;125(10):2342-8. doi: 10.1002/ijc.24642. PMID 19521957
- [Background] Pantuck AJ, Seligson DB, Klatte T, Yu H, Leppert JT, Moore L, O'Toole T, Gibbons J, Belldegrun AS, Figlin RA. Prognostic relevance of the mTOR pathway in renal cell carcinoma: implications for molecular patient selection for targeted therapy. Cancer. 2007 Jun 1;109(11):2257-67. doi: 10.1002/cncr.22677. PMID 17440983
- [Background] Rini BI, Atkins MB. Resistance to targeted therapy in renal-cell carcinoma. Lancet Oncol. 2009 Oct;10(10):992-1000. doi: 10.1016/S1470-2045(09)70240-2. PMID 19796751
- [Background] Wrobel CN, Debnath J, Lin E, Beausoleil S, Roussel MF, Brugge JS. Autocrine CSF-1R activation promotes Src-dependent disruption of mammary epithelial architecture. J Cell Biol. 2004 Apr 26;165(2):263-73. doi: 10.1083/jcb.200309102. PMID 15117969
- [Background] El-Hariry I, Powles T, Lau MR, Sternberg CN, Ravaud A, von der Maase H, Zantl N, Harper P, Rolland F, Audhuy B, Barthel F, Machiels JP, Patel P, Kreuser ED, Hawkins RE. Amplification of epidermal growth factor receptor gene in renal cell carcinoma. Eur J Cancer. 2010 Mar;46(5):859-62. doi: 10.1016/j.ejca.2010.01.011. Epub 2010 Feb 16. PMID 20167476
- [Background] Weber K, Doucet M, Kominsky S. Renal cell carcinoma bone metastasis--elucidating the molecular targets. Cancer Metastasis Rev. 2007 Dec;26(3-4):691-704. doi: 10.1007/s10555-007-9090-y. PMID 17768599
- [Background] Tang SW, Chang WH, Su YC, Chen YC, Lai YH, Wu PT, Hsu CI, Lin WC, Lai MK, Lin JY. MYC pathway is activated in clear cell renal cell carcinoma and essential for proliferation of clear cell renal cell carcinoma cells. Cancer Lett. 2009 Jan 8;273(1):35-43. doi: 10.1016/j.canlet.2008.07.038. Epub 2008 Sep 21. PMID 18809243
- [Background] Thomas RK, Baker AC, Debiasi RM, Winckler W, Laframboise T, Lin WM, Wang M, Feng W, Zander T, MacConaill L, Lee JC, Nicoletti R, Hatton C, Goyette M, Girard L, Majmudar K, Ziaugra L, Wong KK, Gabriel S, Beroukhim R, Peyton M, Barretina J, Dutt A, Emery C, Greulich H, Shah K, Sasaki H, Gazdar A, Minna J, Armstrong SA, Mellinghoff IK, Hodi FS, Dranoff G, Mischel PS, Cloughesy TF, Nelson SF, Liau LM, Mertz K, Rubin MA, Moch H, Loda M, Catalona W, Fletcher J, Signoretti S, Kaye F, Anderson KC, Demetri GD, Dummer R, Wagner S, Herlyn M, Sellers WR, Meyerson M, Garraway LA. High-throughput oncogene mutation profiling in human cancer. Nat Genet. 2007 Mar;39(3):347-51. doi: 10.1038/ng1975. Epub 2007 Feb 11. PMID 17293865
- [Background] MacConaill LE, Campbell CD, Kehoe SM, Bass AJ, Hatton C, Niu L, Davis M, Yao K, Hanna M, Mondal C, Luongo L, Emery CM, Baker AC, Philips J, Goff DJ, Fiorentino M, Rubin MA, Polyak K, Chan J, Wang Y, Fletcher JA, Santagata S, Corso G, Roviello F, Shivdasani R, Kieran MW, Ligon KL, Stiles CD, Hahn WC, Meyerson ML, Garraway LA. Profiling critical cancer gene mutations in clinical tumor samples. PLoS One. 2009 Nov 18;4(11):e7887. doi: 10.1371/journal.pone.0007887. PMID 19924296
- [Background] Broom R, Du H, Clemons M, Eton D, Dranitsaris G, Simmons C, Ooi W, Cella D. Switching breast cancer patients with progressive bone metastases to third-generation bisphosphonates: measuring impact using the Functional Assessment of Cancer Therapy-Bone Pain. J Pain Symptom Manage. 2009 Aug;38(2):244-57. doi: 10.1016/j.jpainsymman.2008.08.005. Epub 2009 Apr 11. PMID 19364633
- [Background] Heng DY, Xie W, Regan MM, Warren MA, Golshayan AR, Sahi C, Eigl BJ, Ruether JD, Cheng T, North S, Venner P, Knox JJ, Chi KN, Kollmannsberger C, McDermott DF, Oh WK, Atkins MB, Bukowski RM, Rini BI, Choueiri TK. Prognostic factors for overall survival in patients with metastatic renal cell carcinoma treated with vascular endothelial growth factor-targeted agents: results from a large, multicenter study. J Clin Oncol. 2009 Dec 1;27(34):5794-9. doi: 10.1200/JCO.2008.21.4809. Epub 2009 Oct 13. PMID 19826129
- [Background] Motzer RJ, Hutson TE, Tomczak P, Michaelson MD, Bukowski RM, Rixe O, Oudard S, Negrier S, Szczylik C, Kim ST, Chen I, Bycott PW, Baum CM, Figlin RA. Sunitinib versus interferon alfa in metastatic renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):115-24. doi: 10.1056/NEJMoa065044. PMID 17215529
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009